CLINICAL TRIAL: NCT04526990
Title: A Global Multicenter, Randomized, Double-blind, Placebo -Controlled, Adaptive Designed Phase Ⅲ Clinical Trial to Evaluate the Efficacy, Safety and Immunogenicity of Ad5-nCoV in Adults 18 Years of Age and Older
Brief Title: Phase III Trial of A COVID-19 Vaccine of Adenovirus Vector in Adults 18 Years Old and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Beijing Institute of Biotechnology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CS-CTP-AD5NCOV-Ⅲ
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: COVID-19; vaccine; Ad5; Safety; Immunogencity; efficacy; adaptive design; SARS-CoV-2; Adenovirus Vector
MeSH Terms: conditions — COVID-19; Alzheimer Disease 5

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 20000 participants, Ad5-nCoV , single dose, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Placebo group (Placebo Comparator): 20000 participants, placebo, single dose, Intramuscular administration
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) — Intramuscular administration
  Arms: Experimental group
Biological: Placebo — Intramuscular administration
  Arms: Placebo group

SUMMARY:
This study is a global multicenter, randomized, double-blind, placebo -controlled, adaptive designed phase Ⅲ clinical trial, in order to evaluate the efficacy, safety and immunogenicity of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) in adults 18 years old and above.

DETAILED DESCRIPTION:
This is a global phase III clinical trial to evaluate efficacy,safety, immuogenicity of Ad5-nCoV manufactured by Cansino and Beijing Institute of Biotechnology in health adults aged 18 years old and above.

The study will be double-blind, placebo-controlled trial with participants randomly allocated 1:1 to placebo and experimental vaccine cohorts.

The immunization schedule is one doses intramuscular injections (deltoid).

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years old and above.
* Participants who are at high risk of SARS-CoV-2 infection.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner/personal doctor and access all medical records when relevant to study procedures.
* Agreement to refrain from blood donation during the study.
* provide written informed consent.

Exclusion Criteria:

* Participation in any other COVID-19 prophylactic drug trials for the duration of the study.
* Participation in SARS-CoV-2 serological surveys where participants are informed of their serostatus for the duration of the study.
* Planned receipt of any vaccine (licensed or investigational), other than the study intervention, within 14 days before and after study vaccination.
* Prior receipt of an investigational or licensed vaccine likely to impact on the interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months prior to the planned administration of the vaccine candidate.
* Planned receipt of any vaccine (licensed or investigational), other than the study intervention, within 14 days before and after study vaccination
* Prior receipt of an investigational or licensed vaccine likely to impact on the interpretation of the trial data (e.g. Adenovirus vectored vaccines, any coronavirus or SARS vaccines)
* Administration of immunoglobulins and/or any blood products within the three months prior to the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state; positive HIV status; asplenia; recurrent severe infections and chronic use.
* History of allergic disease or reactions likely to be exacerbated by any component of Ad5-nCoV
* Any history of angioedema
* Any history of anaphylaxis to any vaccine component
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition likely to affect participation in the study
* Suspected or known current alcohol or drug dependency
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness
* History of laboratory-confirmed COVID-19
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44247 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID-19 cases | day 28 to 12 months post vaccination
  The efficacy of Ad5-nCoV in preventing virologically confirmed (PCR positive) COVID-19 disease
Incidence of SAE | Within 12 months
  Evaluate the incidence of severe adverse events (SAE)

SECONDARY OUTCOMES:
Incidence of severe COVID-19 cases | Day 14 to 12 months post vaccination
  Evaluate the efficacy of Ad5-nCoV in preventing severe COVID-19 disease caused by SARS-CoV-2 infection
Incidence of solicited adverse reactions | Day 0-7 post vaccination
  Incidence of solicited adverse reactions within 7 days after vaccination, in a subset
Incidence of unsolicited adverse events | Day 0-28 post vaccination
  Incidence of unsolicited adverse events within 28 days after vaccination in a subset
Immunogencity of S-RBD IgG antibody (ELISA method) | Day 28 post vaccination
  The seroconversion rate of S-RBD IgG antibody post vaccination
Immunogencity of neutralizing antibody | Day 28 post vaccination
  The seroconversion rate of neutralizing antibody
Cell-mediated immune profile | Day 28 post vaccination
  Number of cell-mediated immune response against SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Halperin, MD, Principal Investigator — Canadian Center for Vaccinology; Fengcai Zhu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention; Joanne M angley, MD, Principal Investigator — Canadian Center for Vaccinology
Locations (73):
- Argentina (12):
  - Fundación Socolinsky Centro de Vacunación Proteger - Recoleta, CABA, Buenos Aires
  - Hospital Pirovano, CABA, Buenos Aires
  - Htal de Alta Complejidad Cuenca Alta Néstor Kirchner, Cañuelas, Buenos Aires
  - Hospital Interzonal de Agudos "San Juan de Dios" de La Plata, La Plata, Buenos Aires
  - Hospital Rossi, La Plata, Buenos Aires
  - Inst. Médico Platense, La Plata, Buenos Aires
  - Instituto de Investigaciones Clínicas, Mar del Plata, Buenos Aires
  - Htal Mariano y Luciano de la Vega, Moreno, Buenos Aires
  - Hospital Houssay, Vicente López, Buenos Aires
  - Hospital Zonal General de Agudos "Cetrangolo", Vicente López, Buenos Aires
  - Instituto Cer, Vicente López, Quilmes
  - Previvax Centro de Vacunación, Córdoba
- Chile (7):
  - Hospital Base de Osorno, Osorno, Los Ríos Region
  - Clinica Alemana de Valdivia Valdivia, Valdivia, Los Ríos Region
  - Clínica Andes Salud Concepción, Concepción, Maule Region
  - Hospital Dr. Hernan Henriquez Aravena Temuco, Temuco, Región de la Araucanía
  - CIMER Centro de Investigaciones Medicas Respiratorias Santiago, Providencia, Santiago Metropolitan
  - Hospital San Borja Arriarán Santiago, Santiago, Santiago Metropolitan
  - Hospital de Puerto Montt Dr. Eduardo Schütz Schoroeder Puerto Montt, Port Montt, X Región de Los Lagos
- Mexico (22):
  - Centro de investigación Médica Aguascalientes (CIMA), Aguascalientes, Aguascalientes
  - Instituto de Servicios de Salud del Estado de Baja California, Mexicali, Baja California Norte
  - Centro de Investigacion Integral MEDIVEST SC, Chihuahua City, Chhihuahia
  - Clinical Research Institute Saltillo SA de CV, Saltillo, Cuahuila
  - Centro de Investigación Clínica del Pacifico S.A. de C.V. (CICPA), Acapulco de Juárez, Guerrero
  - Asociación Mexicana para la investigación clínica (AMIC), Pachuca, Hidalgo
  - Instituto Jaliscience de Metabolismo, S. C., Guadalajara, Jalisco
  - Centro de Investigacion Clinica Chapultepec SA de CV (Hidra), Coyoacán, Mexico City
  - Instituto Mexicano del Seguro Social (IMSS), Cuahtemoc, Mexico City
  - Instuto de Ciencias Médicas y de la Nutrición Salvador Subirán (INCMNSZ), Tlalpan, Mexico City
  - Instituto Nacional de Medicina Genómica, Tlalpan, Mexico City
  - Asociación de investigación pediátrica y adultos (AINPAD), Morelia, Mochoacán de Ocampo
  - JM Research, Cuernavaca, Morelos
  - Hospital Metropolitano "Dr. Bernardo Sepúlveda", San Nicolás de los Garza, Nuevo León
  - Oaxaca site management organization (OSMO), Oaxaca City, Oaxaca
  - Centro de Investigación y Avances Médicos Especializados (CIAME), Cancún, Quintana Roo
  - FAICIC, Veracruz, Veracrua
  - Kohler & Milstein Research, Mérida, Yucatán
  - Instituto de Investigaciones aplicada a las Neurociencias (IIAN), Durango
  - Instituto Nacional de Pediatría (INP), Mexico City
  - PEMEX, Mexico City
  - Administración de Especialistas de Puebla S.C. (UDEP), Puebla City
- Pakistan (5):
  - Shifa International Hospital, Islamabad, Islamabad
  - Shaukat Khanum Memorial Cancer Hospital and Research Centre, Lahore, Punajb
  - University of Health Scinces, Lahore, Lahore, Punjab Province
  - Aga Khan University Hospital, Karachi, Sindh
  - The Indus Hospital, Karachi, Sindh
- Russia (27):
  - Research Center Eco-safety, Saint Petersburg, Sankt-Peterburg
  - OOO Meditsinskie Tekhnologii, Saint Petersburg, Sankt-Peterburg
  - OOO "Baltijskaya Meditsina", Saint Petersburg, Sankt-Peterburg
  - Federal State Budgetary Institution "Scientific Research Institute of Influenza named after A. A. Smorodintsev" of the Ministry of Healthcare of the Russian Federation named after A. A. Smorodintsev" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg, Sankt-Peterburg
  - Saint Petersburg State Budgetary Healthcare Institution "City Polyclinic #106", Saint Petersburg, Sankt-Peterburg
  - Saint-Petersburg State Healthcare Institution "Nikolaev Hospital", Saint Petersburg, Sankt-Peterburg
  - OOO "Piterclinica", Saint Petersburg, Sankt-Peterburg
  - State Budgetary Healthcare Institution of Sverdlovsk Region "Aramil City Hospital", Aramil, Sverdlovsk Oblast
  - Non-state Institution of Healthcare "Road Clinical Hospital at Chelyabinsk station of open corporate society "Russian Railways", Chelyabinsk
  - State Budgetary Educational Institution of Higher Professional Education "Chita State Medical Academy" of the Ministry of Healthcare of the Russian Federation, Chita
  - Federal State Budgetary Institution "Main Military Clinical Hospital n.a. N.N. Burdenko" Ministry of Defense of Russian Federation, Moscow
  - Moscow State Budgetary Healthcare Institution "City Polyclinic #2 of the Moscow City Healthcare Department", Moscow
  - Health Central Clinical Hospital of Russian Academy of Sciences, Moscow
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of Ministry of Healthcare of the Russian Federation (Sechenovsky University), Moscow
  - Private Healthcare Institution "Central Clinical Hospital "RZhD-Medicine", Moscow
  - State Regional Budgetary Healthcare Institution "Murmansk Regional Clinical Hospital n.a.P.A. Bayandin", Murmansk
  - State Regional Autonomous Healthcare Institution "Monchegorsk Central District Hospital", Murmansk
  - Private Healthcare Institution "Clinical Hospital "RZHD-Meditsina" of Nizhniy Novgorod", Nizhny Novgorod
  - "Life Benefits Service, Ltd', Novosibirsk
  - Budgetary Institution of Heathcare of Omsk region "City Clinical Hospital #1 n.a. Kabanova A.N.", Omsk
  - Federal State Budgetary Educational Institution of Higher Education "Perm State Medical University named after E.A. Vagnera" Ministry of Healthcare of Russian Federation, Perm
  - OOO Zvyezdnaya Klinika, Saint Petersburg
  - Limited Liability Company "Hospital "OrKli", Saint Petersburg
  - OOO "Tsentr DNK issledivaniy", Saratov
  - Federal State Budgetary Educational Institution of Higher Education "Saratov State Medical University named after V.I. Razumovsky" the Ministry of Health of the Russian Federation - Clinical hospital n.a. S.R.Mirotvortseva, Saratov
  - OOO "Zdorovye", Tomsk
  - State Autonomous Healthcare Institution of Yaroslavl region "Clinical Emergency Hospital named after N.V. Solovyev", Yaroslavl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halperin SA, Ye L, MacKinnon-Cameron D, Smith B, Cahn PE, Ruiz-Palacios GM, Ikram A, Lanas F, Lourdes Guerrero M, Munoz Navarro SR, Sued O, Lioznov DA, Dzutseva V, Parveen G, Zhu F, Leppan L, Langley JM, Barreto L, Gou J, Zhu T; CanSino COVID-19 Global Efficacy Study Group. Final efficacy analysis, interim safety analysis, and immunogenicity of a single dose of recombinant novel coronavirus vaccine (adenovirus type 5 vector) in adults 18 years and older: an international, multicentre, randomised, double-blinded, placebo-controlled phase 3 trial. Lancet. 2022 Jan 15;399(10321):237-248. doi: 10.1016/S0140-6736(21)02753-7. Epub 2021 Dec 23. PMID 34953526